CLINICAL TRIAL: NCT04203043
Title: Double Blind Randomized Clinical Trial Comparing Pycnogenol Versus Placebo for Pigmentation Prevention After Treatment With Varicose Veins With Foam Sclerotherapy
Brief Title: The Prevstain Trial
Acronym: TPT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, NELSON DE LUCCIA, head of vascular surgery, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08890918.0.0000.0068
Record Dates: First submitted 2019-11-28; First posted 2019-12-18 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pycnogenol oral product to prevent Hyperpigmentation (Active Comparator): Evaluate hyperpigmentation post foam sclerotherapy with placebo versus pycnogenol use
  Interventions: Drug: Pycnogenol Oral Product
- Placebo to prevent hyperpigmentation (Placebo Comparator): Evaluate hyperpigmentation post foam sclerotherapy with placebo versus pycnogenol use
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pycnogenol Oral Product — pycnogenol use to prevent hyper pigmentation after foam sclerotherapy
  Arms: Pycnogenol oral product to prevent Hyperpigmentation
Other: Placebo — Placebo
  Arms: Placebo to prevent hyperpigmentation

SUMMARY:
To evaluate whether oral supplementation with Pycnogenol (Flebon®) can interfere with skin hyperpigmentation after polidocanol foam sclerotherapy in patients with mild to moderate chronic venous insufficiency (CEAP C2 and C3) compared with the use of Placebo.

DETAILED DESCRIPTION:
A randomized double-blind study with research centers in the state of São Paulo (Hospital das Clínicas de São Paulo (HC-SP)) is proposed. Treatment groups: Group 1: Elastic stockings + FlebonGroup 2: Use of elastic socks + Placebo de Flebon.1 Visit 1 - Screening and Selection (D-15) • Evaluation of inclusion and non-inclusion criteria • FICT signature • Clinical evaluation • Aberdeen questionnaire (without schematic design) • Randomization • Dispensation of medication (placebo and Pycnogenol) • Dismissal of use diary 2. Visit 02 D0 - Initiation of treatment (+/- 2 days) • Performing the procedure by Sclerotherapy • Record of adverse events • Pre-sclerotherapy photographic record • Clinical evaluation • investigational product (placebo and Pycnogenol) • Dismissal of new use diary (elastic stockings and investigational product) • Withdrawal criteria • Visit 03 - D7 - Return of 7 days (+/- 2 days) • Evaluation of withdrawal criteria • Evaluated adherence to treatment by use diary • Return of control (eventual drainage) • Record of adverse events • Clinical evaluationVisit 04 - D30 - Return 30 days after visit 2 (+/- 2 days) • Treatment adherence assessment by use diary • Photographic control I • Hyperpigmentation scale • Pigment size assessment, if any • Record of adverse events • Assessment of withdrawal criteria • Assessment clinical • Investigational Product Dispensation (Placebo and Pycnogenol) • New Usage Diary DispensationView 05- D60 - Return 60 Days After Sight 3 (+/- 2 days) • Usage Diary Treatment Adherence Assessment • Photographic Control II • Hyperpigmentation Scale • Pigment size assessment, if any • Record of adverse events • Assessment of withdrawal criteria • Assessment • Dispensation of medication (placebo and Pycnogenol) • Dispensation of new use diaryVisit 06 -D90 - Return 90 days after sight 04 (+/- 2 days) • Evaluation of treatment adherence by use diary • Evaluation of criteria • Photographic control III •Pigment size assessment, if any • Aberdeen questionnaire application (without schematic drawing) • Medication suspension • Hyperpigmentation scale • Adverse event recording • Research participant satisfaction rating • Clinical assessmentPhotographic recording of the legs will be performed before 30, 60 and 90 days in 03 (three) incidences and evaluated by 01 blind observer. The photographic records will be made by camera following the same parameters, namely: 60 cm distance to 50 cm from the ground, not using flash, with artificial lighting (ceiling light), without zoom. All generated images will be archived in JPEG (Joint Photographic File Format) format. Images must be downloaded within 5 days of photographic registration and inserted into All images should be encoded as follows: IDENTIFICATION OF PARTICIPANTS + DATE OF PHOTOGRAPH REGISTRATION CO (00/00/0000) + VISIT. In addition, a sticker with the research participant's initials and date of photograph registration should be visible to the image. The blinded study medium will evaluate all photographs at the end of the study, making a comparison between them to inform the presence and the evolution of hyperpigmentation due to foam sclerotherapy, when they occur.For this, the Torok Hyperpigmentation Scale will be applied at D 30, D 60 and D90.

ELIGIBILITY:
Inclusion Criteria:

* Female participants, non-pregnant, aged ≥18 years.
* Phototype Fitzpatrick II to IV
* Participant with mild to moderate chronic venous insufficiency (classification C2 and C3 of the clinical criterion CEAP classification).
* Participant who underwent treatment of the great saphenous vein
* and. Indication for performing lower limb sclerotherapy followed by elastopression for 7 days.
* With indication for procedure by 1% polidocanol sclerotherapy
* Demonstrate understanding of procedures, study restrictions and willingness to participate as evidenced by written informed consent and attendance of all scheduled visits
* Good overall mental and health with, in the opinion of the investigator or medically qualified designee, no clinically significant and relevant abnormalities in medical history or upon physical examination.
* Exclusion Criteria:
* The. Pregnancy or intention to become pregnant during the study or breastfeeding women.
* Any history of significant dermatological conditions or diseases or medical conditions known to alter skin appearance or physiological response (eg, diabetes, heart failure, hypothyroidism, or hyperthyroidism), which could, in the opinion of the Investigator, prevent and / or interfere with the assessment of the reaction of the test site.
* Active acne (local or widespread) that may interfere with study results.
* Participants currently using any medication, which, in the opinion of the investigator, may affect the evaluation of the study product or subject the participant to excessive risk.
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs and corticosteroids up to 2 weeks before the screening visit.
* Oral or topical treatment with vitamin A or retinoic acid and / or its derivatives up to 1 month before the screening visit.
* Have participated in any clinical study within the last 12 months prior to the start of the study;
* Any clinical and / or laboratory alteration that, in the Investigator's opinion, may interfere with the participant's safety.
* Use of anticoagulant or antiplatelet agent
* BMI greater than 40 kg / m² Uncontrolled diabetes or hypertension
* Recent thrombosis (less than 6 months from inclusion)
* no Participants with a history of polyamide or elastane allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2020-02-28 (Estimated); Primary Completion 2020-03-28 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
photographic evaluation of the presence or absence of skin hyperpigmentation after foam sclerotherapy | 90 days
  To evaluate the impact of Pycnogenol (Flebon®) use on skin hyperpigmentation after sclerotherapy procedure in relation to placebo group, according to the presence or absence of hyperpigmentation.Hyperpigmentation will be assessed through standardized photographs taken by the study researchers and evaluated by a blinded dermatologist in the study. The answer will be dichotomous, yes or no.

SECONDARY OUTCOMES:
The use of Pycnogenol (Flebon®) triggers change cutaneous pigmentation; | 90 days
  The degree of pigmentation involvement will be assessed using the Hyperpigmentation Scale (Torok) by a blinded dermatologist in the study after 30, 60 and 90 days of treatment.
The use of Pycnogenol (Flebon®) triggers a change skin pigmentation. | 90 days
  The size of the pigmentation will be evaluated by the use of a conventional standardized ruler, considering the largest pigmentation axis, verified in millimeters, after 30, 60 and 90 days of treatment.
The use of Pycnogenol (Flebon®) change the signs and symptoms of chronic venous insufficiency by applying a CVI-specific quality of life questionnaire. | 90 days
  Improvement of signs and symptoms of chronic venous insufficiency will be assessed by applying the Aberdeen questionnaire (without schematic design) at baseline and after 90 days of treatment.
the degree of patient satisfaction with the use of Pycnogenol (Flebon®) regarding the skin aspect of the region submitted to the procedure; | 90 days
  The degree of patient satisfaction will be made subjectively by the study participants through a scale from 0 to 6, 0 being totally dissatisfied and 6 fully satisfied after 90 days of treatment.
pycnogenol side effects | 90 days
  report any type of adverse event